CLINICAL TRIAL: NCT05441904
Title: A Phase I, Two-part, Single and Optional Multiple Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of 500 and 750 mg PXL770 in Healthy Subjects
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics of PXL770 in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Poxel SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PXL770-009
Record Dates: First submitted 2022-06-22; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: NASH - Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 2-chloro-3-(1-hydroxy-5,6,7,8-tetrahydronaphthalen-2-yl)-6-oxo-5-phenyl-7H-thieno)(2,3-b)pyridin-4-olate potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PXL770 500 and 750 mg (Experimental): Each subject received 1 dose of PXL770 at 500 mg and 1 dose at 750 mg
  Interventions: Drug: PXL770

INTERVENTIONS:
Drug: PXL770 — A single dose of 500 and 750 mg was administered to each subject.

SUMMARY:
The study was planned in 2 parts: Parts A and B. In Part A, we tested 2 single doses of the study medicine in healthy volunteers: 500 mg and 750 mg. Part B was an optional part to test once-daily doses of the study medicine in healthy volunteers. We aimed to assess the safety, tolerability find out the side effects and blood levels of the PXL770.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female healthy volunteer.
2. Aged 18-55 years.
3. A body mass index in the range 18.5-29.9.
4. Body weight at least 50 kg.
5. Sufficient intelligence to understand the nature of the trial and any hazards of participating in it. Ability to communicate satisfactorily with the investigator and to participate in, and comply with the requirements of, the entire trial.
6. Willingness to give written consent to participate after reading the information and consent form, and after having the opportunity to discuss the trial with the investigator or their delegate.
7. Agree to follow the contraception requirements of the trial.
8. Agree not to donate blood or blood products during the study and for up to 3 months after the administration of the trial medication.
9. Willingness to give written consent
10. Registered with a General Practitioner in the UK.

Exclusion Criteria:

1. Woman who is pregnant or lactating, or pre-menopausal woman who is sexually active and not using a reliable method of contraception.
2. Clinically relevant abnormal history, physical findings, ECG, or laboratory values at the pre-trial screening assessment that could interfere with the objectives of the trial or the safety of the volunteer.
3. Presence of acute or chronic illness or history of chronic illness sufficient to invalidate the volunteer's participation in the trial or make it unnecessarily hazardous.
4. Estimated glomerular filtration rate at screening < 90 mL/min/1.73 m2 (estimated using the method established by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI]).
5. History of drug-induced Torsade de Pointes, or known risk factors for Torsade de Points (heart failure, hypokalemia, short QT syndrome, family history of long QT Syndrome, or QTcF > 450 msec (men) or > 470 msec (women). Triplicate QTcF measurements will be taken at screening, and a mean QTcF value higher than 450 msec (men) or 470 msec (women) will lead to exclusion. A repeat (in triplicate) is allowed on one occasion for determination of eligibility.
6. Impaired endocrine, thyroid, hepatic, respiratory or renal function, diabetes mellitus, coronary heart disease, or history of any psychotic mental illness.
7. Surgery (stomach bypass) or medical condition that might affect absorption of medicines.
8. Presence or history of severe adverse reaction to any drug or a history of sensitivity to PXL770, or its excipients.
9. Presence or history of anaphylactic or anaphylactoid reaction or food allergy.
10. Use of a prescription medicine (except oral contraceptives or hormone replacement therapy in women), over-the-counter medicine with the exception of acetaminophen (paracetamol), dietary supplement or herbal remedy during the 14 days before the first dose of trial medication.
11. Receipt of an investigational product (including prescription medicines) as part of another clinical trial within the 3 months before first admission to this study; in the follow-up period of another clinical trial at the time of screening for this study.
12. Have previously taken PXL770 in another clinical trial.
13. Presence or history of drug or alcohol abuse, or intake of more than 14 units of alcohol weekly, or more than 5 cigarettes, 1 cigar or pipe (about ¼ ounce tobacco) daily.
14. Regular consumption of more than 5 cups of caffeinated drinks (or equivalent) daily.
15. Blood pressure and heart rate in supine position at the screening examination outside the ranges: blood pressure 90-140 mm Hg systolic, 40-90 mm Hg diastolic; heart rate 40-100 beats/min. Borderline values (ie values that are within 5 mm Hg for blood pressure or 5 beats/min for heart rate) will be repeated in triplicate. Subjects can be included if the repeat value is within range or still borderline but deemed not clinically significant by the investigator.
16. Vegetarians or vegans, or unwilling to eat up to two breakfasts including bacon.
17. Possibility that the volunteer will not cooperate with the requirements of the protocol.
18. Evidence of drug abuse on urine testing, or positive urine alcohol test.
19. Positive test for hepatitis B, hepatitis C or human immunodeficiency virus (HIV). Participants with positive hepatitis C antibody due to prior resolved disease can be included if the hepatitis C ribonucleic acid (RNA) test is obtained and the result is negative.
20. Loss of more than 550 mL blood during the 3 months before the trial.
21. Objection by General Practitioner to volunteer in the trial.
22. Involved in the planning or conduct of the study at Poxel S.A. or HMR.
23. Considered a vulnerable person (a prisoner on probation, for example).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Cmax | Blood samples for assay of PXL770 will be taken at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours after each dose.
  maximum concentration
AUC | Blood samples for assay of PXL770 will be taken at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours after each dose.
  area under the curve
t1/2 | Blood samples for assay of PXL770 will be taken at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours after each dose.
  half-life
tmax | Blood samples for assay of PXL770 will be taken at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours after each dose.
  time to reach maximum concentration
MRT | Blood samples for assay of PXL770 will be taken at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours after each dose.
  mean residence time
CL/F | Blood samples for assay of PXL770 will be taken at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours after each dose.
  apparent clearance
Vz/F | Blood samples for assay of PXL770 will be taken at pre-dose and at 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72, 96, 120 and 144 hours after each dose.
  volume of distribution

SECONDARY OUTCOMES:
AE | Safety monitoring will be done from the date of signature of the ICF until the end of the study, assessed up to 5 weeks.
  Adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- HMR, London, NW10, United Kingdom

IPD SHARING:
Plan to Share IPD: No